CLINICAL TRIAL: NCT06507579
Title: Prospective Observational Study on the Efficacy and Safety of Hydra Transcatheter Aortic Valve
Brief Title: Hydra Registry - UK
Status: Recruiting | Type: Observational
Sponsor: Sahajanand Medical Technologies Limited (Industry)
Collaborators: Psephos Biomedica (Unknown)
Responsible Party: Sponsor
Other Study IDs: HYD/SHEFFIELD-001/2023
Record Dates: First submitted 2024-07-03; First posted 2024-07-18 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Valve Stenosis, TAVI, Hydra
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe aortic valve stenosis: Hydra transcatheter aortic valve (THV) series
  Interventions: Device: Hydra transcatheter aortic valve (THV) series

INTERVENTIONS:
Device: Hydra transcatheter aortic valve (THV) series — The Hydra device consists of a self-expanding nitinol frame and three bovine pericardial leaflets in supra-annular position.

SUMMARY:
The study will evaluate the efficacy and safety of transcatheter aortic valve implantation (TAVI) using the Hydra transcatheter aortic heart valve (THV) series, in patients with severe aortic stenosis up to 1-year after the procedure. This will include an evaluation of the preservation of coronary access post implant by attempting to selectively engage both the right and left coronary arteries through standardised angiographic views.

The study will also examine the utility of 72 hours of post discharge remote ambulatory continuous electrocardiogram (ECG) monitoring using the novel Checkpoint Cardio System where it is clinically appropriate.

DETAILED DESCRIPTION:
This is a prospective, observational, multi-centre study. The aim of this study is to collect clinical, procedural, and follow-up data in order to evaluate the efficacy and safety of the Hydra THV series (Vascular Innovations Co. Ltd., Nonthaburi, Thailand).

Additionally, the study will conduct the following evaluation:

1. The remote ambulatory cardiac monitoring (rACM) using the Checkpoint Cardio System, consisting of 72 hours of continuous electrocardiogram (ECG) monitoring, will be evaluated post hospital discharge where it is clinically appropriate.
2. Coronary access will be evaluated immediately post-TAVI by attempting to selectively engage both the right and left coronary arteries through standardised angiographic views. This will be done in a sub-set of patients who are either known to have coronary artery disease, did not have coronary angiogram prior to TAVI or where it is felt to be clinically appropriate for other reasons post implant.

Following discharge, clinical follow-ups are scheduled at 45 days (±14 days), and 1-year (±30 days).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe aortic stenosis eligible for transfemoral TAVI procedure as per local Heart Team evaluation
2. Full understanding and willing to provide informed consent to study enrolment
3. Age ≥ 18 years

Exclusion Criteria:

1. Contraindications to TAVI (e.g., anatomically phenotypes, intracardiac mass, thrombus, vegetation, endocarditis)
2. Refusal to provide informed consent to study enrolment
3. Patients with severe aorta or peripheral artery disease precluding transfemoral approach of TAVI
4. Patients with significant calcification of the aortic annulus and in the Left Ventricular Outflow Tract (LVOT), or/and excess calcium within each cusp, or those who are deemed unsuitable for the Hydra THV series based on the clinical judgment of the Investigator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or Female
Study Population: Patient with severe aortic valve stenosis
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-07-11 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint | 45 days
  Early safety as defined by VARC-3 as composite of:
  * Freedom from all-cause mortality;
  * Freedom from all stroke;
  * Freedom from VARC 3 type 3-4 bleeding;
  * Freedom from major vascular, access-related, or cardiac structural complication;
  * Freedom from acute kidney injury stage 3 or 4;
  * Freedom from moderate or severe aortic regurgitation;
  * Freedom from new permanent pacemaker due to procedure-related conduction abnormalities;
  * Freedom from surgery or intervention related to the device.
Primary performance endpoint | 45 days
  Device success as defined by VARC-3 as composite of:
  * Technical success;
  * Freedom from mortality;
  * Freedom from surgery or intervention related to the device or to a major vascular or access related or cardiac structural complication;
  * Intended performance of the valve (mean gradient <20mmHg, peak velocity <3 m/s, Doppler velocity index ≥0.25, and less than moderate aortic regurgitation).

SECONDARY OUTCOMES:
Technical success | Immediately after the procedure
  As per VARC-3 defined criteria
Cardiovascular mortality | 45 days, and 1-year
All-cause mortality | 45 days, and 1-year
All stroke | 45 days, and 1-year
Disabling stroke | 45 days, and 1-year
Myocardial infarction | 45 days, and 1-year
Major vascular complication | 45 days
Acute kidney injury | 45 days
New permanent pacemaker implantation due to procedure related conduction abnormalities | 45 days, and 1-year
New-onset atrial fibrillation | 45 days, and 1-year
Coronary artery obstruction requiring intervention | 45 days, and 1-year
Re-hospitalization for procedure- or valve-related causes | 45 days, and 1-year
Mean aortic valve gradient | 45 days, and 1-year
Effective Orifice Area (EOA) | 45 days, and 1-year
Paravalvular leak | 45 days, and 1-year
New York Heart Association (NYHA) functional class | 45 days, and 1-year
Change in quality-of-life score assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | 45 days, and 1-year
  Assessed by the Kansas City Cardiomyopathy Questionnaire (KCCQ-12)
Bioprosthetic Valve Failure (BVF), defined as valve-related mortality or aortic valve re-operation/re-intervention, or stage 3 haemodynamic severe structural valve deterioration | 45 days, and 1-year
Bioprosthetic valve dysfunction (BVD), defined as structural valve deterioration, non-structural valve deterioration, clinical valve thrombosis, infective endocarditis | 45 days, and 1-year
Stroke or peripheral embolism (presumably valve-related, after ruling out other non-valve aetiologies) | 45 days, and 1-year
VARC-3 Type 3-4 bleeding secondary to or exacerbated by antiplatelet or anticoagulant agents used specifically for valve-related concerns (e.g., clinically apparent leaflet thrombosis) | 45 days, and 1-year
Significant arrhythmias on rACM that would potentially lead to permanent pacemaker implantation (PPMI) | 72 hours post hospital discharge
Ability to selectively engage and obtain diagnostic epicardial coronary angiography images from the right and left coronary ostia | Immediately post-TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Javaid Iqbal, MRCP, PhD, Principal Investigator — Northern General Hospital, Sheffield Teaching Hospitals NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Northern General Hospital, Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, Yorkshire
  - Royal Victoria Hospital, Belfast
  - Royal Papworth, Cambridge
  - Castle Hill Hull, Cottingham

IPD SHARING:
Plan to Share IPD: No